CLINICAL TRIAL: NCT01966614
Title: Randomized, Double-Blind, Vehicle-Controlled, Multicenter Safety and Efficacy Study of a Single Intraprostatic Treatment of PRX302 for Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostatic Hyperplasia (The PLUS 1 Trial)
Brief Title: Randomized, Double-Blind, Vehicle-Controlled, Multicenter Safety and Efficacy Study of Intraprostatic PRX302 for LUTS BPH
Acronym: PLUS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRX302-3-01
Record Dates: First submitted 2013-10-14; First posted 2013-10-21 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; BPH; Enlarged prostate; Lower urinary tract symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — PRX302

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRX302 (Experimental): PRX302 injection
  Interventions: Drug: PRX302
- Placebo (Placebo Comparator): Placebo (Vehicle-only injection)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRX302 — Single intraprostatic bilateral injection at a dose of 0.6 µg/g
  Other Names: topsalysin
  Arms: PRX302
Other: Placebo — Single intraprostatic bilateral injection of vehicle only
  Other Names: Vehicle-only
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a single treatment of PRX302 for the treatment of Benign Prostatic Hyperplasia (BPH) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Lower Urinary Tract Symptoms (LUTS) attributable to BPH for ≥6 months
* IPSS ≥15
* Maximum urine flow (Qmax) of 5 - 15 mL/sec
* Prostate volume of 30 - 100 mL as determined by TRUS
* Serum prostate-specific antigen (PSA) values <10 ng/mL
* Post-void residual (PVR) <= 200 mL

Exclusion Criteria:

* Inability to void ≥125 mL urine
* Prior surgery/MIST for BPH
* Presence of or history of certain conditions that could interfere with study results or endanger subject
* Use of certain prescribed medications that could interfere with study results

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | Week 52
  International Prostate Symptom Score (IPSS) total score change from baseline over 52 weeks.

SECONDARY OUTCOMES:
Efficacy | Week 52
  Qmax change from baseline over 52 weeks.
Efficacy | Week 52
  IPSS total score change from baseline at each individual post-baseline timepoint.
Efficacy | Week 52
  Qmax change from baseline at each individual post-baseline timepoint.
Efficacy | Week 52
  IPSS "responders" at each individual post-baseline timepoint.
Efficacy | Week 52
  Qmax "responders" at each individual post-baseline timepoint.
Efficacy | Week 52
  Proportion of patients who receive rescue therapy.
Efficacy | Week 52
  Time to onset of rescue therapy.
Efficacy | Week 52
  Incidence rate for episodes of urinary retention.
Efficacy | Week 52
  Transition Zone (TZ) prostate volume change from baseline as measured by transrectal ultrasound (TRUS) at each individual post-baseline timepoint.
Efficacy | Week 52
  Total prostate volume (PV) change from baseline as measured by TRUS at each individual post-baseline timepoint.
Safety | Week 52
  Treatment-emergent adverse events (TEAEs).
Safety | Week 52
  Episodes of acute urinary retention as determined by the independent Adjudication Panel.
Safety | Week 52
  Assessment of sexual function for men who are sexually active using the International Index of Erectile Function - Erectile Function (IIEF-EF) and the Male Sexual Health Questionnaire© short form for ejaculatory dysfunction (MSHQ-EjD).
Safety | Week 52
  Physical examinations.
Safety | Week 52
  Vital signs.
Safety | Week 6
  Electrocardiograms (ECGs).
Safety | Week 52
  Laboratory parameters, consisting of chemistry panel, complete blood count (CBC), and urinalysis.
Safety | Week 52
  Measurement of anti-PRX302 antibodies (APA).
Safety | Week 52
  Serum concentration of PRX302 only if clinically indicated by an event such as suspected systemic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Yocum, MD, Study Director — Sophiris Bio Corp
Locations (65):
- United States (43):
  - Huntsville, Alabama
  - Anchorage, Alaska
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - San Diego, California
  - Tarzana, California
  - Denver, Colorado
  - Middlebury, Connecticut
  - Aventura, Florida
  - Coral Gables, Florida
  - Pompano Beach, Florida
  - St. Petersburg, Florida
  - Wellington, Florida
  - Coeur d'Alene, Idaho
  - Meridian, Idaho
  - Springfield, Illinois
  - Jeffersonville, Indiana
  - West Des Moines, Iowa
  - Baltimore, Maryland
  - Greenbelt, Maryland
  - Towson, Maryland
  - Brookline, Massachusetts
  - Missoula, Montana
  - Mount Laurel, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - New York, New York
  - Newburgh, New York
  - Poughkeepsie, New York
  - The Bronx, New York
  - Concord, North Carolina
  - Raleigh, North Carolina
  - Bala-Cynwyd, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Greer, South Carolina
  - Myrtle Beach, South Carolina
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Burien, Washington
- Australia (4):
  - Daw Park, South Australia
  - Woodville South, South Australia
  - Mentone, Victoria
  - Parkville, Victoria
- Canada (3):
  - Brampton, Ontario
  - Kitchener, Ontario
  - Oakville, Ontario
- New Zealand (3):
  - Whau Valley, Whangarei
  - Christchurch
  - Tauranga
- Russia (5):
  - Ivanovo
  - Moscow
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
- Ukraine (7):
  - Chernihiv
  - Chernivtsi
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Zaporizhzhya